CLINICAL TRIAL: NCT05844514
Title: The COlorectal BReath Analysis (COBRA2) Study: Non-invasive Breath Testing to Detect Colorectal Cancer
Brief Title: COlorectal BReath Analysis (COBRA2)
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Chelsea and Westminster NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other); Royal Marsden NHS Foundation Trust (Other); London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 17SM3783 - SA 04
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer
Keywords: Volatile organic compounds; Breath analysis; Volatolomics; Mass spectrometry
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Breath Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group - 470 patients: Symptomatic patients who are attending a planned colonoscopy referred under the suspected lower GI cancer pathway. Any patient who is found to have histologically-proven CRC on colonoscopy will be analysed as part of the CRC group.
  Interventions: Diagnostic Test: Breath test
- CRC group - 250 patients: Patients who either have a confirmed diagnosis of colorectal adenocarcinoma according to a biopsy, or who are due to undergo surgical resection for suspected CRC (with histological confirmation to follow within three months).
  Interventions: Diagnostic Test: Breath test

INTERVENTIONS:
Diagnostic Test: Breath test — Patients must be fasted for a minimum of 4-6 hours prior to breath sample collection. For patients undergoing colonoscopy or surgery, breath samples must be obtained prior to patients receiving bowel preparation in either outpatient clinic or pre-assessment clinic.

SUMMARY:
Colorectal cancer (CRC) is the second most common cause of cancer death in the United Kingdom, with approximately 17,000 deaths per year. The five-year survival rate from CRC is only 10% when discovered at a late stage, but exceeds 90% if diagnosed early. Symptoms related to CRC can be non-specific, therefore the decision to refer for a colonoscopy can be challenging.

There is a clear need to improve earlier detection of CRC so that patients with CRC can be identified earlier and faster, enabling them to start treatment more quickly.

The study team is developing a non-invasive breath test that detects small molecules called volatile organic compounds (VOCs) that are specific to CRC. For patients with non-specific symptoms, this test would help GPs to identify those patients that may have underlying CRC, who would benefit from referral for specialised CRC tests.

DETAILED DESCRIPTION:
The COBRA1 study initially assessed VOCs in CRC and identified a list of 14 VOC biomarkers for CRC and provided a detection model with an area under the receiver operating characteristic curve of 0.91, sensitivity of 83% and specificity of 88% in symptomatic patients.

COBRA2 aims to develop and validate the clinical prediction model (CPM) in the detection of CRC based on the breath test. An exploratory comparison between the breath test and faecal immunochemical test (FIT) will also be carried out to assess whether combining both tests improves diagnostic performance.

Methods: COBRA2 is be a prospective, multicentre validation study. The study team are recruiting the following patients:

The following groups of patients are being recruited:

i) Control group: symptomatic patients who are attending a planned colonoscopy referred under the suspected lower GI cancer pathway. Any patient who is found to have histologically-proven CRC on colonoscopy will be analysed as part of the CRC group.

ii) CRC group: patients who either have a confirmed diagnosis of colorectal adenocarcinoma according to a biopsy, or who are due to undergo surgical resection for suspected CRC (with histological confirmation to follow within three months).

Target recruitment is 720 patients (470 controls, 250 CRC), aiming for 576 patients (376 controls, 200 CRC) with reliable and complete data. Participants are required to maintain a clear fluid diet for a minimum of 4-6 hours prior to sampling and should not have received bowel preparation. Participants will be asked to provide breath samples by exhaling into single-use breath collection bags and breath will be transferred using a precision pump onto thermal desorption (TD) tubes. Breath samples will be analysed with gas chromatography-mass spectrometry in accordance with existing quality control processes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years referred from primary care with symptoms of suspected CRC.
* Patients with histologically confirmed colorectal adenocarcinoma (stages I-IV) who are treatment naïve (CRC group).

Exclusion Criteria - patients with any of the following will not be eligible for inclusion:

* Previous surgery altering the anatomy of the lower GI tract (e.g., hemicolectomy, anterior resection).
* Previous treatment (neoadjuvant chemotherapy or radiotherapy or immunotherapy) for CRC.
* Received bowel preparation for their colonoscopy procedure.
* History of any other cancer within three years.
* Unable or unwilling to provide informed written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seen in a hospital (secondary or tertiary level care) setting
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Validation and further discovery of VOC biomarkers for CRC. | 24 months
  GC-MS will be used to confirm the presence of certain CRC-associated VOCs in order to develop the detection model.

SECONDARY OUTCOMES:
Exploratory comparison between the breath test and FIT. | 24 months
  Assessment of the performance of combining both the breath test and FIT to detect CRC.

CONTACTS AND LOCATIONS:
Overall Officials: Professor George B Hanna, PhD FRCS, Principal Investigator — Imperial College London
Locations (5):
- United Kingdom (5):
  - Chelsea and Westminster Hospital, London
  - Royal Marsden Hospital, London
  - St Mark's Hospital, London
  - St Mary's Hospital, London
  - West Middlesex University Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fadel MG, Murray J, Woodfield G, Belluomo I, Laponogov I, Parker A, Converso V, Ellis JK, Wheatstone P, Hepburn J, Groves C, Monahan K, Saunders BP, Spanel P, Veselkov K, Cross AJ, Kontovounisios C, Sharples LD, Hanna GB; COBRA2 Collaborators. Non-invasive breath testing to detect colorectal cancer: protocol for a multicentre, case-control development and validation study (COBRA2 study). BMC Cancer. 2025 Jul 29;25(1):1230. doi: 10.1186/s12885-025-14520-2. PMID 40731329